CLINICAL TRIAL: NCT05027100
Title: One Arm, Exploratory Study of Tislelizumab Combined With Anlotinib and 2-cycle Irinotecan Monotherapy as Second Treatment of Small Cell Lung Cancer
Brief Title: Tislelizumab Combined With Anlotinib and 2-cycles Irinotecan as Second Line Treatment of SCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haibo Zhang (Other)
Responsible Party: Sponsor-Investigator, Haibo Zhang, Chief Physician, Guangzhou University of Traditional Chinese Medicine
Organization: Guangzhou University of Traditional Chinese Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.0/20201227
Record Dates: First submitted 2021-08-22; First posted 2021-08-30 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Safety and effectiveness of tislelizumab combined with anlotinib and 2-cycle irinotecan monotherapy as second line treatment of small cell lung cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exploratory research (Experimental): Anlotinib 10mg QD with 2W stop 1W tiselizumab injection 200mg Q3W Irinotecan (2 cycles) 100mg/m2,d1,d8,Q3W
  Interventions: Drug: Anlotinib Tislelizumab Irinotecan

INTERVENTIONS:
Drug: Anlotinib Tislelizumab Irinotecan — Anlotinib 10mg QD 2W stop 1W Tislelizumab injection200mg Q3W Irinotecan (2 cycles) 100mg/m2,d1,d8,Q3W

SUMMARY:
SCLC has short doubling time, high proliferation rate and early widespread metastasis. Most patients with SCLC have hematogenous metastasis. SCLC is highly sensitive to initial chemoradiotherapy, but the recurrence rate is high. The strategy for local limited SCLC patients was chemotherapy plus chest radiotherapy; In patients with extensive stage SCLC, first-line platinum-based chemotherapy has been established as the standard treatment for patients with small cell lung cancer (SCLC) with better results. Although the initial response to chemotherapy is high, it is easy to relapse and develop drug resistance.

In second-line therapy, the single-agent activity of multiple chemotherapy agents has been demonstrated, but a higher incidence of grade 3-4 hematological adverse events In the Passion study published by Wang Jie et al. [10], the efficacy and safety of the antiangiogenic drug apatinib combined with carrizumab in the second-line treatment of small cell lung cancer were investigated. A total of 59 patients were enrolled in the study. Of the 47 patients in the extended phase, the confirmed ORR was 34.0% (95%CI 20.9-49.3), with a median PFS of 3.6 months and a median OS of 8.4 months In patients with platinum sensitivity and platinum resistance, ORR was 37.5% vs 32.3%, MPFS was 3.6m vs 2.7m, and MOS was 9.6m vs 8.0m. Grade 3 treatment-related adverse events (TRAEs) occurred in 43 of the 59 patients (72.9%), and 5 patients (8.5%) were discontinued due to TRAEs. The combination regimen showed potential antitumor activity in both platinum-sensitive and platinum-resistant cases.

The research and exploration of small cell lung cancer can learn from the research idea in the field of non-small cell lung cancer. The Checkmate9LA study reported in 2020ASCO [11] investigated the safety and efficacy of Nivolumab+2 cycle chemotherapy in first-line treatment of non-small cell lung cancer with negative driver gene. The MOS in the immunization combination group was significantly better than that in the chemotherapy group (15.6 months vs. 10.9 months, HR 0.66), and the 1-year survival rate was 63% vs. 47%, respectively. The ORR in the immunization combination group was also improved (38% vs. 25%), and the MDOR was 11.3m vs. 5.6m, which was tolerable in terms of safety. The incidence of grade 3-4 treatment-associated AE was 47% in the immune-combined group and 38% in the chemotherapy group. From the perspective of mechanism, chemotherapy can enhance the immunogenicity of tumor cells, damage the immune cell inhibitory activity, which can induce tumor cell apoptosis, expression of MHC class 1 molecules increases and mature dendritic cells to promote the immune response, in the design, add 2 cycles of chemotherapy short-term intensive treatment, make up the immune short board, For example, the early onset of slow and immune characteristic events such as large tumor load, pseudo progression, hyperrogression and other problems, to achieve the optimization and upgrading of the scheme.

Based on Rationale 307, Tislelizumab was approved on January 12, 2021 for first-line treatment in combination with paclitaxel and carboplatin in patients with locally advanced or metastatic squamous non-small cell lung cancer. t the same time, Tislelizumab initial efficacy in patients with extensive small-cell lung cancr.Rational-206 study is a phase Ⅱ multi-cohort study of Tislelizumab combined with first-line platinum-containing chemotherapy in patients with advanced lung cancer in China. The MPFS in the SCLC cohort was about 7 months, and the MOS reached 15.6 months.

Based on the above studies and data, in the second-line treatment of SCLC, anti-vascular targeted drugs combined with chemotherapy can obtain a certain survival benefit, especially for patients with sensitive recurrence, and the benefit is more significant. he immune checkpoint inhibitors have gradually emerged in the second-line and later treatment of SCLC, but the single drug effect has not been a great breakthrough; a small molecule antiangiogenic targeted drug in China, Anlotinib has obtained third-line and later indications of SCLC through ALTER1202 data, and has been included in the 2019 CSCO Guidelines for the Diagnosis and Treatment of Primary Lung Cancer. t the same time, it is similar to the Checkmate9LA study regimen, combined with two cycles of chemotherapy, to improve the short-term efficacy. Therefore, Anlotinib combined with Tislelizumab, a PD-1 inhibitor, and 2 cycles of Irinotecan monotherapy were tried in second-line SCLC, with the hope of breaking through the difficulties of high recurrence rate and rapid disease progression of existing second-line SCLC chemotherapy, regardless of platinum-sensitive recurrence or platinum-resistant recurrence, and providing more options for SCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteered to participate in this study and signed the informed consent, with good compliance and follow-up;
2. Male or female patients aged between 18 and 75 years;
3. Patients with extensive small-cell lung cancer diagnosed by pathology, who have received first-line chemotherapy/PD-L1(CSCO rocommended standard therapy ) and failed treatment, and who have measurable target lesions; Definition of treatment failure: disease progression or intolerance during or after chemotherapy treatment for who have previously received concurrent chemoradiotherapy or adjuvant chemotherapy, if recurrence/metastasis occurs within 6 months after the end of the last treatment, the original treatment plan is defined as the subject's first-line treatment plan.
4. The interval between the time of disease progression and the end of the last systemic chemotherapy was less than 6 months;
5. Life expectancy of at least 3 months, ECOG score: 0-1;
6. The main organs are functioning normally

Exclusion criteria:

1. Patients with previous use of anlotinib capsules or other antiangiogenic drugs;
2. Previous use of tislelizumab injection other anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies, as well as any other antibody or drug therapy targeting T cell co-stimulatory or checkpoint pathways, such as ICOs or agonists (such as CD40, CD137, GITR, Ox40, etc.);
3. Patients who have previously used Irinotecan injection or other camptothecin drugs
4. Patients who have received two or more platinum-containing two-drug chemotherapy (adjuvant chemotherapy relapse time within 6 months is counted as first-line chemotherapy);
5. Imaging (CT or MRI) showed obvious pulmonary cavitary tumor;
6. History and complications
7. Unacceptable toxicity after prior anti-PD-L1 treatment is defined as follows:

A. Grade ≥ 3 AE associated with anti-PD-L1 therapy that does not respond to standard therapy and requires treatment termination.

B. Grade ≥ 2 imAE associated with anti-PD-L1 therapy, unless AE is restored or well controlled after discontinuation of anti-PD-L1 therapy and/or steroid therapy, except for prior colitis, encephalitis, myocarditis, hepatitis, uveitis, and lung inflammation.

C. Any grade of CNS or ocular AE associated with anti-PD -L1. Note: Patients with prior endocrine AE are allowed to be enrolled if they remain stable and asymptomatic after appropriate alternative therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
ORR(Investigator-assessed) | up to 48months
  Tumor remission is revaluted by investigator according to RECIST v 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 48months
  The time from enrollment to (for any reason) progress disease
overall survival (OS) | up to 48months
  The time from enrollment to (for any reason) death.
(Disease control rate assessed by investigators) DCR (CR+PR+SD) | up to 48months
  The time from the first recorded objective tumor response (CR or PRorSD) to objective
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Adverse events will be assessed during the period of 2cycles of treatment (21 days for each cycle), since the date of randomization. Adverse events will be recorded once any side effect happens.
  Treatment-emergent adverse events is defined as any adverse events happened after randomization. The severity is validated using NCI-CTCAE V4.03.

CONTACTS AND LOCATIONS:
Overall Officials: haibo zhang, Professor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No